CLINICAL TRIAL: NCT00381966
Title: A Pilot Study of Robotic Template Guidance for Needle Placement in Transperineal Prostate Brachytherapy
Brief Title: Study of Robotic Template Guidance for Needle Placement in Transperineal Prostate Brachytherapy
Acronym: J0511
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: J0511; 5R44CA088139-04 (NIH); 05-03-28-03 (Other: JHM IRB); SBIR Ph1/Ph2 (Other: other)
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Results first posted 2018-06-29 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- Robotic placement device (Experimental): The intervention involves use of a robotic template to assist in placement of needles for prostate brachytherapy.
  Interventions: Device: robotic placement device

INTERVENTIONS:
Device: robotic placement device — this device is a robotic arm that utilizes a template as a guidance system to precisely inplant radioactive brachytherapy seeds directly to the prostate.
  Other Names: template guided robotic placement tool

SUMMARY:
This is a study that will try see if a device can help to better guide the needle that places prostate cancer treatment.

DETAILED DESCRIPTION:
Section 1- Background:

Adenocarcinoma of the prostate will affect over 220,900 U.S. males this year, making it the most prevalent cancer in the nation.1 Prostate specific antigen (PSA) is a very useful tumor marker in early detection of this malignancy, as well as a reliable marker for control after definitive therapy with either surgery or irradiation. Widespread use of prostate-specific antigen (PSA) screening has resulted in approximately 45% of patients being detected with early stage disease. For this group of patients, brachytherapy or implantation of radioactive sources into the prostate is a treatment option that has risen dramatically in use over the last several years due to its effectiveness and convenience.

The use of brachytherapy or implantation of radioactive sources into the prostate for adenocarcinoma has advantages over external beam radiation in that a very high dose can be delivered to the tumor while limiting the doses to the surrounding normal tissue (i.e., bowel and bladder). It is well established that outcomes after treatment with brachytherapy are critically related to the technical quality of source placement within the gland. A spatially desirable placement of the radioactive sources with achievement of optimum dose distributions within the prostate is key to the success of brachytherapy with regard to both killing tumor as well as minimizing toxicity.

The development of transrectal ultrasound (TRUS) of the prostate, with the ability to map the prostate in several planes, as well as the associated development of trans-perineal implantation of the prostate, has allowed the development of the modern prostate implantation method. Ultrasound images are taken before or during the implant procedure, and a source distribution plan is developed that optimizes dose to the prostatic tissues while sparing the urethra and rectum. Needles are placed into the prostate via a transperineal template, and the sources are placed into the prostate according to the source distribution plan.

Currently, the template utilized for needle guidance is limited to 0.5 centimeter x-axis and y-axis grid spacing, limiting the ability of the needle positions to conform to the shape of the prostate, which is spherical (Fig 1). The most commonly utilized method of dosimetric planning involves placing needles around the periphery of the prostate capsule, in order to best cover potential microscopic extracapsular extension as well as to avoid the dose sensitive urethra which runs through the center. The grid arrangement of the current template limits the ability of these needle positions to best approximate the external contour of the prostate (Fig 2). Also, placement of sources in the most posterior row adjacent to rectum is critical. Sources too close to rectum may cause increased risk of rectal bleeding, whereas source too far from the capsule may result in risk of underdosing disease in that area. Greater freedom in needle positioning would allow for more optimum placement of sources.

Figure 1. Transperineal template device 3 Figure 2. Grid positions available with traditional template (white dot grid on screen). Prostate outline is seen on the image.

Researchers in the Johns Hopkins University (JHU) School of Engineering have developed a robotic needle positioning device which will allow greater flexibility in choosing needle positions for prostate brachytherapy. The device consists of a motor attached to a needle guidance hole. The entire apparatus attaches to the ultrasound 'stepper' device similar to the standard transperineal template. For each needle position, the motor moves to the predetermined location and the physician places the needle through the hole. Visual verification of acceptable needle position is performed by viewing the needle on the real-time ultrasound. A secondary means of verification will be the use of an Optical Tracking device, which will verify needle orientation and position prior to insertion. Rather than having the probe positioned at the desired endpoint of the needle insertion within the prostate, the ultrasound unit will be mechanically coupled with the needle (via the optical tracking system) as it is being inserted, such that the needle tip will be continuously visualized as it is progressing into the prostate.

Another problem frequently encountered in brachytherapy is pubic arch interference. Given the proximity of the prostate to the pubic arch, the anterior aspect of the prostate often abuts this structure. If pubic arch curves posteriorly around the inferior aspect of the prostate, then access to the anterior prostate with transperineal needles is limited. Some patients may not be eligible for brachytherapy due to this problem with their anatomy.

This device will allow for angulation of needles such that pubic arch interference may be circumvented by inserting more posteriorly and then angling the needle anteriorly such that the pubic arch is not in the needle path as it travels toward the anterior prostate.

We will use the Computerized Medical Systems (CMS) Interplant system software (St Louis, MO), which has the capability of calculating treatment plans using sources off of the usual template grid positions.

Section 2 -Objectives:

This will be a feasibility trial of a therapeutic device. The purpose of the study is to demonstrate the clinical feasibility of using the needle positioner device in a cohort of 5 patients. This will involve demonstrating the feasibility of using the system in an actual operating room environment and determining acceptable positioning effectiveness by assessing needle position during insertion on the live ultrasound image, as well as by using an optical tracking device.

Section 3- Study Population:

The eligible population will be patients with a diagnosis of adenocarcinoma of the prostate who are seen in consultation at the Johns Hopkins Hospital.

Patient accrual (5 patients) is expected to complete within 3-5 months.

Section 4 - Protocol Design:

This will be a feasibility study with a cohort of 5 patients. 4.1. Subject Identification: Patient confidentiality will be maintained in accordance with Health Information Portability and Accountability Act (HIPAA) guidelines. All participants must sign an informed consent that will describe the objectives of the study and potential risks. All patient data reported on the case reports forms will be identified by the patient's initials and study code number only. Patients shall not be identified by name. This should serve to protect the confidentiality of subjects enrolled on the trial. Clinical data and records for all subjects studied including history and physical

findings, laboratory data, and results of interventions are to be maintained by the investigators in a secure, locked location. Computerized data will require password authorization(s) for access.

4.2. Description of the Recruitment Process: Potential subjects will be identified at the time of consultation in the Department of Radiation Oncology by Dr. Song. All patients meeting above stated eligibility criteria will be offered participation in the study by the consulting physician.

4.3. Description of the Informed Consent Process: Only physicians who are investigators on this project will perform the informed consent interview. The informed consent interview will take place prior to the day the patient is to be treated to ensure that the patient has adequate time to discuss the research project with family, friends, and/or other Health Care providers. During the informed consent interview the interviewer (investigator) will take as much time as needed to ensure that the potential subject understands the research project and also clearly understands that he does not have to participate in this project to receive his cancer treatment at Johns Hopkins. If the patient decides to enroll into the research project he will sign three copies of the informed consent form. One will be for his own records, one will be kept in the Clinical Research Office at Johns Hopkins, and the third one will be kept in his medical records.

4.4. Subject Assignment: Five patients will be enrolled onto the trial. 4.5. PATIENT ASSESSMENTS Assessments Pre-Study Entry Post Brachytherapy Month 3 (+/- 4 weeks) History/physical Exam Xa X KPS Xa PSA Xa X Chest X-ray Xa Xb CT of pelvis Xa Xb Ultrasound volume Xa Bone scan (if clinically indicated) Xa

1. within 6 weeks prior to day 1 of brachytherapy
2. up to 1 day post brachytherapy RADIATION THERAPY AND RESEARCH INTERVENTIONS The patient population who will be offered this protocol are those who are currently offered brachytherapy as standard treatment at our institution. The clinical protocol will not affect what patients experience during the procedure.

Implant procedure As is our routine, within the week prior to implantation the patient will undergo a transrectal ultrasound study to determine the volume of the prostate and estimate the number of sources required. A preliminary implant plan will be developed based on the pre-operative ultrasound.

On the day of implantation, the patient will be brought into the operating room and 'timeout' performed. He will be placed in dorsal lithotomy position after anesthetic (either general or spinal) is administered. A foley catheter will be placed into the urethra. Ultrasound images will be acquired and a dosimetric plan developed based on the intraoperative ultrasound. Computerized dosimetric algorithms are used to assist the physician in creating a plan which adequately treats the prostate while minimizing dose to urethra and rectum.

Given that the needle positioner device will allow an infinite number of positions rather than being limited to predetermined holes, the source placement will be planned by the physician with this in mind. Sources are placed with immediate feedback from software as to dosimetric ramifications on normal tissues and prostate coverage. If a source position does not correspond to the usual template grid, the software allows the user to 'drag' the closest grid needle position to the desired location.

Instead of a standard template with pre-drilled holes mounted on the ultrasound support mechanism, the needle positioner device will be attached to the stepper unit. Needles are inserted through the needle positioner, through the perineum and into the prostate, using positions dictated by the dosimetric plan. Ultrasound guidance is used to visualize and guide the needle placement. An optical tracking system (Northern Digital Inc, Waterloo Canada) with measured accuracy of 0.1 millimeter, will be used to track the needle position and angle prior to insertion into tissue.

The correctness of the needle position produced by the needle positioning device (NPD) will be ascertained at two levels, before committing the needle to insertion and during insertion. The tracker will be placed in the field of surgery. The tracker will be calibrated to the coordinate space of the template. Then the template is removed and the NPD is placed. The tracker will be calibrated to the coordinate space of the NPD too. Assuming that the tracker does not move during the procedure, this establishes a direct spatial co-registration between the coordinate space of a template and NPD. At any time during the procedure, the current position of the NPD and needle guide can be reported to the responsible physician in template coordinates. Thus the physician will compare the current needle position (reported in template space) to the desired needle position determined by the treatment plan (also in template space). In case of any discrepancy between the reported and desired needle positions, the NPD is removed and replaced by the template, and the procedure continues without delay.

During needle insertion, the ultrasound will move in synch with the needle insertion (via optical tracking and motorized control of the ultrasound probe) in order to allow constant visualization of the needle tip during insertion. The depth of insertion of the ultrasound probe is limited by the stepper unit which it is attached to. After each needle insertion, C-arm fluoroscopy is briefly used to assess and confirm the positioning, and a Mick applicator (Mick Radio-Nuclear Instruments, Mount Vernon NY) will be used to place sources into the prostate via the needle. Following source placement the needle is removed, the needle positioner moves to the next needle position, and the procedure is repeated until all sources have been placed. After all sources are placed, a final set of fluoroscopic images is taken for confirmation and documentation.

When using the standard transperineal template, the template is calibrated to the ultrasound probe prior to the implant procedure by using a phantom, such that the grid on the template accurately correlates to the grid as seen on ultrasound. However, during the actual procedure it is not uncommon for the needle position as visualized on ultrasound to be slightly displaced from the predicted location. This is due to needle bending from tissue forces during insertion. When this occurs the physician removes the needle and repeats the insertion with mild force on the needle at the point of tissue entry in order to achieve the desired position. The needle guide may also be recalibrated if successive needle attempts show consistent deviation in one direction, which is indicative of slight errors in calibration. This is not an unusual finding in typical practice.

For purposes of this study, the needle positioning system will also be calibrated prior to each implant. However, if during the procedure the physician finds that the needle positioner is inaccurate in a non- systematic fashion (not related to slight calibration error) relative to the intended position, the system can be quickly replaced by the standard template during the procedure, since it mounts to the stepper in identical fashion.

Other treatment Patients who have either Gleason score of 7 or PSA 10-20 will be treated with external beam radiation in addition to brachytherapy in accordance with our usual practice.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are unchanged from our standard criteria for brachytherapy eligibility:

* Histologically confirmed, locally confined adenocarcinoma of the prostate
* Clinical stages T1b - T2b
* PSA of less than 20 ng/mL
* Combined Gleason score 7 or less, with no individual Gleason score of 5
* The patient has decided to undergo brachytherapy at the Johns Hopkins Hospital as treatment choice for his prostate cancer.
* Karnofsky Performance Status (KPS) > 70
* Prostate volume by TRUS < 50 cc
* International Prostate symptom score (IPSS) must be 18 or less
* Signed study-specific consent form prior to registration

Exclusion Criteria:

* Stage T1a, or T3 or greater disease.
* Clinical or Pathological Lymph node involvement (N1).
* Evidence of distant metastases (M1).
* Radical surgery for carcinoma of the prostate.
* Previous Chemotherapy or pelvic radiation therapy
* Previous transurethral resection of the prostate (TURP)
* Significant obstructive symptoms (IPSS greater than 18)
* Hip prosthesis.
* Anatomic or medical condition (such as prior abdominal-perineal resection or anal stricture) which would preclude the use of TRUS

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Song, M.D., Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Robotic Placement Device
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Robotic Placement Device
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Positioning Effectiveness as Determined by Confirmatory Measurements of Robotic Movements
Description: Confirmatory measurements of robotic movements was assessed using infrared tracking to calculate mean error in millimeters.
Time Frame: at time of intervention
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Robotic Placement Device
Number analyzed (Participants) | 5
millimeters | 0.489 (0.328)

2. Primary Outcome: Utility of the Needle Position Device: Number of Adjustments Possible Out of Adjustments Attempted
Description: Utility was demonstrated in terms of fine adjustments (≤ 2 mm) and adjustments >2mm in needle positioning, being possible when tissue deflection was encountered.
Time Frame: at time of intervention
Measure: Count of Units; unit: Number of Adjustments
Units Other Than Participants: Number of Adjustments
Arm/Group | Robotic Placement Device
Number analyzed (Participants) | 5
Number analyzed (Number of Adjustments) | 54
Number of Adjustments
  Adjustments ≤ 2 mm | 18
  Adjustments > 2 mm | 36

ADVERSE EVENTS:
Description: Adverse events were not collected or assessed as part of the study.
Arm/Group | Robotic Placement Device
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No